CLINICAL TRIAL: NCT02026427
Title: The Incidence of Urinary Retention in Orthopedic Patients Under Spinal Anesthesia
Brief Title: Urinary Retention in Orthopedic Patients
Acronym: UriRet
Status: Completed | Type: Observational
Sponsor: Military Institute od Medicine National Research Institute (Other)
Responsible Party: Principal Investigator, Dariusz Tomaszewski, MD, PhD, Military Institute od Medicine National Research Institute
Other Study IDs: 06101968-1
Record Dates: First submitted 2013-12-31; First posted 2014-01-03 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-08

CONDITIONS: Urinary Retention; Orthopedic Patients; Spinal Anesthesia
MeSH Terms: conditions — Urinary Retention

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Drotaverine: 40 mg of drotaverine hydrochloride administered intramuscularly just after the proper level of spinal anesthesia was achieved.
- Control: Without intramuscular administration of drotaverine hydrochloride.

SUMMARY:
The participants were hospitalized in Orthopedic and Traumatology Departments in Military Institute of Medicine, Warsaw, Poland.

The inclusion criteria were (1) age to 40 year-old, (2) no history of urologic problems, and (3) surgery under spinal anesthesia. All the patients where (1) opioids were administered during the surgery, (2) general anesthesia was necessary, and (3) the urinary bladder catheterization was perform during the surgery were excluded from the study.

The participants were randomly divided into the study and control groups. No oral premedication was administered. All the patients were asked to empty their urinary bladders before arrival to the operating theatre. When the standard monitoring (continuous electrocardiogram, noninvasive blood pressure, pulse oximetry) was started, intravenous premedication with midazolam was administered and lumbar spinal anesthesia with hyperbaric 0.5% solution of bupivacaine hydrochloride was performed.

In the study group, but not in the the control one, the 40 mg of drotaverine hydrochloride was administered intramuscularly. The decresed intravascular volume was corrected with cristalloids. During the surgery the adequate, not deeper than II grade according to Ramsay scale, level of sedationt was obtained with midazolam and/or propofol. All the participants received a questionaire in which we asked the questions about (1) the duration of anesthesia, (2) the time of micturition, (3) the time when discomfort or pain appeared in the lower abdomen, (4) the incidence of the urinary bladder catheterization and time to catheterization. On the next day after the surgery the questionaires were collected. In cases, when the patient's dischaged from the hospital was planned during the weekend, he or she was asked to pass on the questionaire to the nurses.

ELIGIBILITY:
Inclusion Criteria:

* age below 40 y.o.,
* surgery under spinal anesthesia,
* no previous history of urological problems.

Exclusion Criteria:

* opioid administration during surgery,
* need for urinary bladder catheterization during surgery,
* conversion to general anesthesia.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients scheduled for orthopedic surgery under spinal anesthesia.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2010-08; Primary Completion 2014-06 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
time to micturition | first 24 hours after spinal anesthesia
  Time (in minutes) from the administration of spinal anesthesia to spontaneous micturition.

SECONDARY OUTCOMES:
urinary bladder catheterization | first 24 hours after spinal anesthesia
  1. the need of urinary bladder catheterization, and
  2. time from administration of spinal anesthesia to catheterization

CONTACTS AND LOCATIONS:
Locations (1):
- Military Institute of Medicine, Warsaw, Poland

REFERENCES:
- [Derived] Tomaszewski D, Balkota M. Intramuscular Administration of Drotaverine Hydrochloride Decreases Both Incidence of Urinary Retention and Time to Micturition in Orthopedic Patients under Spinal Anesthesia: A Single Blinded Randomized Study. Biomed Res Int. 2015;2015:926953. doi: 10.1155/2015/926953. Epub 2015 Jun 21. PMID 26185766